CLINICAL TRIAL: NCT01275534
Title: Patient Reported Outcomes in View of Symptom Experience of Late Effects and Self-management After Haematopoietic Stem Cell Transplantation - A Mixed Methods Study
Brief Title: Symptom Experience and Self-management After Haematopoietic Stem Cell Transplantation
Acronym: PROVIVO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 264-10
Record Dates: First submitted 2011-01-03; First posted 2011-01-12 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Hematologic Neoplasms
Keywords: Stem cell transplantation; Symptom experience; Late effects; Self-management
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In the study PROVIVO, a patient reported outcome instrument consisting of items from the PRO-CTCAE item bank measuring symptom experience of long-term survivors after allogeneic hematopoietic stem cell transplantation (SCT) will be developed. The instrument development is based on cognitive patient interviews, a survey of hematology experts and a literature review. In a subsequent cross-sectional study phase, the instrument will be validated in a sample of 300 allogeneic stem cell recipients and by the use of additional self report instruments it will be possible to explore how subjective symptom experience, problems in self-management and presence of late effects are connected.

DETAILED DESCRIPTION:
Long-term survivors after allogeneic SCT are presumably at a life-long increased risk for developing various adverse side effects; also termed 'late effects'. Late effects may appear months or years after treatment has ended, can persist chronically and may be experienced as rather distressing and burdensome. Since most late effects are only experienced subjectively in the form of physical and mental symptoms and are seldom captured during objective clinician-based evaluations, using self-report instruments is important for the early detection, management and alleviation of these symptoms. The collection of self-report data in studies and clinical practice is strongly recommended by the National Cancer Institute (NCI): they developed a Patient-Reported Outcomes bank based on the well established Common Terminology Criteria for Adverse Events (PRO-CTCAE).

Besides managing symptoms associated with late-effects, patients with SCT are also requested to manage their emotions associated with having a chronic illness, their new life roles in order to have a meaningful, fulfilling life, and their medical regimen, in view of taking medications, smoking cessation, regularly exercising and monitoring for signs of infection. However, evidence investigating the prevalence of problems related to these complex set of self-management tasks is scarce.

Aims:

* To translate the PRO-CTCAE items into German in a culturally-sensitive way and to develop the content of a self-report instrument measuring symptom experience after allogeneic SCT
* To validate the newly developed scale and assess its psychometric properties
* To examine self reported symptom experience and objective measured late effects in 300 adult survivors ≥ 1 year after SCT
* To describe self-management behaviours in 300 adult survivors ≥ 1 year after SCT
* To assess the relationship between symptom experience and objective burden of late effects, survivors' perception of late effects and self-management in view of managing emotions, managing new life roles and managing medical and health tasks in 300 adult survivors ≥ 1 year after allogeneic SCT

ELIGIBILITY:
Inclusion Criteria:

* Having received allogeneic SCT for haematological disease
* ≥ 1 year of follow-up experience after treatment
* Ability to understand and read German and having signed the written informed consent

Exclusion Criteria:

* Patients with psychiatric illness that in the opinion of physicians prevent them from participating
* Visual and/or hearing impairment which hinders participation in an interview/fill-out a questionnaire
* Being illiterate
* Actual acute care hospitalization stay at interview date
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long-term survivors after allogeneic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Symptom experience | single measuring point at ≥ 1 year after HSCT
  Patient reported symptom experience using items of the PRO-CTCAE

SECONDARY OUTCOMES:
Perception of late effects | single measuring point at ≥ 1 year after HSCT
  Brief Illness Perception Questionnaire
Self-management behaviors | single measuring point at ≥ 1 year after HSCT
  Patient reported self-management behaviors measured by single items
Self-management in view of medical and health tasks, emotional and role tasks | single measuring point at ≥ 1 year after HSCT
  Patient reported self-management behaviors using single items and the Hospital Anxiety and Depression Scale
Objective late effects | single measuring point at ≥ 1 year after HSCT
  Physician graded late effects using the CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sabina De Geest, PhD, Principal Investigator — University of Basel
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Kirsch M, Mitchell SA, Dobbels F, Stussi G, Basch E, Halter JP, De Geest S. Linguistic and content validation of a German-language PRO-CTCAE-based patient-reported outcomes instrument to evaluate the late effect symptom experience after allogeneic hematopoietic stem cell transplantation. Eur J Oncol Nurs. 2015 Feb;19(1):66-74. doi: 10.1016/j.ejon.2014.07.007. Epub 2014 Sep 1. PMID 25190633